CLINICAL TRIAL: NCT03598049
Title: Assessment of Dental Implants Placed in Posterior Maxillary Ridge Using Densah Burs Versus Standard Drills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira khaled ahmed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 47820
Record Dates: First submitted 2018-06-29; First posted 2018-07-26 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Implant Site Reaction
Keywords: Implants; Stability; Bone loss; Success
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- densah burs drilling group (Experimental): implant osteotomy site drilling using the densah burs osseo densification drills
  Interventions: Device: densah burs osseo densification drills
- surgical burs drilling group (Active Comparator): implant osteotomy site drilling using conventional surgical burs drilling
  Interventions: Device: conventional surgical burs drilling

INTERVENTIONS:
Device: densah burs osseo densification drills — osseo densification of the alveolar bone in maxillary posterior ridge during implant placement
  Arms: densah burs drilling group
Device: conventional surgical burs drilling — conventional implant osteotomy site drilling with implant surgical kit
  Arms: surgical burs drilling group

SUMMARY:
comparing the drilling technique of using densah burs osseo densification drills in posterior maxilla with the normal surgical kit drilling

DETAILED DESCRIPTION:
the densification of bone using the densah burs are thought to be improving the bone quality surrounding the implants thus increasing the primary stability and decreasing the marginal bone loss surrounding the implants comparing to the normal drilling techniques using the conventional implant drilling kit

ELIGIBILITY:
Inclusion Criteria:

* Patients with partially edentulous in the posterior area of the maxilla, with a residual ridge that allowed insertion of ≤3.5 width implants.
* Both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement

Exclusion Criteria:

* Sinus pathology.
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site
* Immunodeficiency pathology, bruxism, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
implant stability | at the time of surgery
  measurement of implant stability using the ostell

SECONDARY OUTCOMES:
Marginal bone loss | 3 month
  measurement of the bone level surrounding the implant using cone beam CT

OTHER OUTCOMES:
patient satisfaction | 3 month
  patient satisfaction questionnaire